CLINICAL TRIAL: NCT01775891
Title: Efficacy of Pilsicainide After Radiofrequency Ablation of Paroxysmal Atrial Fibrillation Compared With Other Class IC Anti-arrhythmic Drugs
Brief Title: Efficacy of Pilsicainide After Radiofrequency Ablation of Paroxysmal Atrial Fibrillation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Korea University (Other)
Responsible Party: Principal Investigator, Young-Hoon Kim, M.D. PhD, Korea University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PIL245
Record Dates: First submitted 2013-01-23; First posted 2013-01-25 (Estimated); Last update posted 2013-02-26 (Estimated); Status verified 2013-02

CONDITIONS: Paroxysmal Atrial Fibrillation
Keywords: pilsicainide; class IC antiarrhythmic drug; paroxysmal atrial fibrillation; catheter ablation
MeSH Terms: conditions — Atrial Fibrillation | interventions — pilsicainide; Flecainide; Propafenone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- pilsicainide (Active Comparator): The dose of pilsicainide will be 50mg tid PO. Pilsicainide will be started on the night of the ablation for a duration of at least 3 months. Physicians were encouraged to stop the drugs following the 3 months treatment if possible.
  Interventions: Drug: pilsicainide; Drug: other class IC antiarrhythmic drug
- other class IC antiarrhythmic drug (Placebo Comparator): Other class IC antiarrhythmic drug that they had been taking before catheter ablation will be administrated.(flecainide 100mg bid PO or propafenone 225mg tid) Antiarrhythmic drug will be started on the night of the ablation for a duration of at least 3 months. Physicians were encouraged to stop the drugs following the 3 months treatment if possible.
  Interventions: Drug: pilsicainide; Drug: other class IC antiarrhythmic drug

INTERVENTIONS:
Drug: pilsicainide — The dose of pilsicainide will be 50mg tid PO. Pilsicainide will be started on the night of the ablation for a duration of at least 3 months. Physicians were encouraged to stop the drugs following the 3 months treatment if possible.
  Other Names: Pilsicainide (Sunrhythm®) Daiichi Sankyo
Drug: other class IC antiarrhythmic drug — Other class IC antiarrhythmic drug that they had been taking before catheter ablation will be administrated.(flecainide 100mg bid PO or propafenone 225mg tid) Antiarrhythmic drug will be started on the night of the ablation for a duration of at least 3 months. Physicians were encouraged to stop the drugs following the 3 months treatment if possible.
  Other Names: flecainide 100mg bid PO or propafenone 225mg tid

SUMMARY:
Investigators hypothesized that the use of Pilsicainide after radiofrequency ablation of AF could reduce the incidence of recurrence of atrial arrhythmia during follow up compared with other class IC antiarrhythmic drugs.

DETAILED DESCRIPTION:
Catheter ablation has become an integral part of the management of atrial fibrillation (AF), when a strategy to preserve normal sinus rhythm is required. However, recurrence of atrial arrhythmias is common after AF ablation. In order to prevent these arrhythmia recurrences, antiarrhythmic drugs (AADs) are often resumed empirically after AF ablation. Previously a prospective randomized trial demonstrated that the treatment with AADs during the first 6-weeks after AF ablation reduced the incidence of clinically significant atrial arrhythmias and need for cardioversion or hospitalization for arrhythmia management.

Pilsicainide is a class IC antiarrhythmic drug originally developed in Japan, which has a pure sodium channel blocking action with slow recovery pharmacokinetics. Its mechanism of action appears to provide new insight into the pharmacological conversion of AF.

In experimental studies, pilsicainide has a potent depressant effect on intra-atrial conduction and a prolonging effect on the atrial effective refractory period (ERP). Theoretically the suppression of conduction velocity minimizes the prolongation of wavelength induced by the increase in the ERP and may thus serve to allow the continuation of multiple re-entrant wavelets. Iwasa et al demonstrated that pilsicainide was more effective at terminating vagally induced AF than propafenone, despite the greater effect of propafenone on wavelength, suggesting that suppression of conduction velocity may play an important role in terminating AF. Moreover, Wijffels et al reported that the pharmacological cardioversion of AF cannot be explained by the prolongation of wavelength.

The effects of a single oral treatment of pilsicainide were compared with that of a disopyramide infusion in a multicentre trial. Seventy two patients with symptomatic paroxysmal AF were randomised to receive either a single oral dose of pilsicainide (100-150mg) or an infusion of disopyramide (2 mg/kg; maximum dose = 100mg). In the pilsicainide group, the cumulative percentage of conversion to sinus rhythm within 120 minutes was high as disopyramide (73% vs 56%). Moreover, the conversion time of pilsicainide is shorter than that of other class IC antiarrhythmics, including flecainide and propafenone, in patients with recent-onset AF. This seems likely to be due to the favorable pharmacokinetics of pilsicainide, including its rapid absorption from the gastrointestinal tract, the absence of changes from a first-pass effect, and a short elimination half-life.

In the case of an unsuccessful ablation for AF, AADs that were ineffective before the ablation are sometimes effective. The effects and mechanisms of hybrid therapy with pilsicainide and PV isolation for AF have been assessed. Seventy four patients with paroxysmal AF in whom pilsicainide was ineffective underwent PV isolation. A second PV isolation was performed in 31 patients among 42 recurred patients (57%). Pilsicainide was re-administered in recurred patients even after the second session. Amng 21 patients with recurrence of AF, pilsicainide and eliminated AF in 11 patients (success with hybrid therapy was 86%).

In patients with paroxysmal AF, pilsicainide significantly prolonged the ERP of the distal pulmonary vein (PV), PV-left atrium (LA) junction and LA, and the conduction time from the distal PV to the PV-LA junction. In some patients, PV-LA conduction block has been observed just before pilsicainide-induced termination of AF; this isolation of the PV may provide a new insight into the mechanism of pharmacological conversion of AF. Hybrid therapy with pilsicainide and PV isolation (by radiofrequency catheter ablation) appears to be an effective therapeutic approach for AF. The pharmacological PV isolation by pilsicainide and its suppression of focal discharges from atrial tissue may prevent the development of AF after unsuccessful ablation. These mechanism makes it suitable for hybrid therapy with catheter ablation of the PVs.

Therefore investigators hypothesized that the use of Pilsicainide after radiofrequency ablation of AF could reduce the incidence of recurrence of atrial arrhythmia during follow up compared with other AADs. Furthermore, we seek to identify whether there are clinical predictors of AF recurrence at 1-year follow-up and the relationship of early recurrence during blanking period and recurrence during 1-year follow up.

ELIGIBILITY:
Inclusion Criteria:

* patients with drug-refractory paroxysmal atrial fibrillation who requires catheter ablation
* patients who are aged 18-80 and agree with this study

Exclusion Criteria:

* patients who do not agree with this study
* patients with a history of catheter ablatio or surgery for atrial fibrillation
* patients who experienced side effects of pilsicainide before
* patients who has galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption
* patients who has congestive heart failure with ejection fraction<40% or decompensated heart failure
* patients with significant coronary artery disease, liver/renal disease
* patients who has other kinds of arrhythmic which requires active treatment
* contraindication to warfarin therapy
* life expectancy <1 year]
* pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Estimated)
Dates: Start 2012-07; Primary Completion 2015-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
freedom from recurrence of any atrial arrhythmia within 1 year | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Young-Hoon Kim, MD., PhD, Principal Investigator — Arrhythmia center, Anam hospital, Korea university
Locations (1):
- Arrhythmia center, Anam Hospital, Korea University, Seoul, South Korea